CLINICAL TRIAL: NCT02211092
Title: Development and Pilot Testing of a Home-Based Physical Activity Intervention for Family Caregivers of People With Advanced Cancer
Brief Title: Feasibility Study of a Home-based Physical Activity Intervention for Family Caregivers of People With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jamie Penner, RN, PhD(c), Nursing Doctoral Candidate, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-129; 003208 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Self Care; Family Caregivers
Keywords: Family Caregivers; Advanced Cancer; Palliative Care; Support; Self Care; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity intervention (Experimental): A 12 week individually tailored home-based physical activity program with goal-setting, a physical activity self-monitoring technique, and weekly telephone calls provided by the intervener for coaching and support.
  Interventions: Behavioral: Physical activity intervention
- Usual care (Other): Access to usual community resources but no active lifestyle coaching.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Physical activity intervention — A 12 week individually tailored home-based physical activity program with goal-setting, a physical activity self-monitoring technique, and weekly telephone calls provided by the intervener for coaching and support.
  Arms: Physical activity intervention
Other: Usual care — Access to usual community resources but no active lifestyle coaching.
  Arms: Usual care

SUMMARY:
The purpose of this study is to develop an individually tailored home-based physical activity intervention for family caregivers of people with advanced cancer and assess the feasibility of a future randomized controlled trial (RCT) to test the effects of this intervention.

DETAILED DESCRIPTION:
Families play an essential role in the care of people with advanced cancer and usually undertake caregiving responsibilities for patients at home. While caregiving is often rewarding, the physical and emotional demands of caregiving have significant impacts on caregivers' health, including a wide range of emotional responses and high levels of fatigue. Caregivers' own health is important and their ability to continue to provide care also necessitates that their self-care needs are met. However, few supportive interventions have been developed specifically to address these needs. One way of doing so may be increasing physical activity. The physical and psychological benefits of physical activity are well documented. A lifestyle approach to physical activity can be tailored to the needs, preferences, and circumstances of the individual and is therefore a logical way to address some of the self-care needs of caregivers within the context of their personal caregiving situation. The main objectives of this pilot study are to develop an individually tailored home-based physical activity intervention for family caregivers of people with advanced cancer and assess the feasibility of a future randomized controlled trial to test the effect of this intervention on caregivers' positive and negative affect, fatigue, and overall self-rated health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to speak and read English
* involved in the care of a person with advanced cancer (stage III or IV) at home

Exclusion Criteria:

* already participating in physical activity more than three days a week and 30 minutes or more per session as assessed by self-report
* a current mental illness that has been treated with medication for <8 weeks or that the caregiver intends to initiate medication for during the period of the intervention
* any major physical health problem that would prevent caregivers from participating in the intervention as assessed by the Physical Activity Readiness Questionnaire (PAR-Q)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | 9 months of running feasibility trial
  Frequency counts of the number of participants recruited from each of the recruitment sites will be conducted and the overall rate of recruitment will be calculated.
  This criterion for advancing to a full RCT will be met if the estimated sample size required for a full RCT can likely be recruited in 2 years.
Number of participants who drop out | 9 months of running feasibility trial
  Frequency counts for the number of participants who drop out of both the experimental and control group will be conducted and the percentage rate of attrition in each group will be calculated.
  This criterion for advancing to a full RCT will be met if less than 30% of participants dropped out of the experimental or control group.
Number of items complete on the outcome questionnaires | Baseline, 6, 9, and 12 weeks
  To assess acceptability of outcome questionnaires and feasibility of data collection procedures for a full RCT, descriptive statistics (frequency counts) of complete versus incomplete items as well as the expected versus actual completion dates will be conducted at baseline, and week 6, 9, and 12 for both the experimental and control group on the following outcome measures: Positive and Negative Affect Schedule (PANAS); Lee Fatigue Scale (LFS); General Self-Rated Health question.
  This criterion for advancing to a full RCT will be met if less than 10% of items on each of the questionnaires are missing and less than 10% of participants are missing any one item on each of the questionnaires.
Rate of adherence to individual physical activity plans | 12 weeks
  The number of weeks that participants were able to engage in physical activity levels at or above their retrospective baseline physical activity level in relation to the number of weeks that they were in the study will be calculated. Rate of adherence will be calculated for individual participants and the mean and median rate of adherence will be calculated for the experimental group. The proportion of participants that were able to engage in physical activity at or above their retrospective baseline level of physical activity 0-25%, 26-50%, 51-75%, and 76-100% of the time will be calculated.
  Qualitative data will also be collected and analyzed to explore what factors influence adherence to the individual physical activity plans.
  This criterion for advancing to a full RCT will be met if the rate of adherence to the individual PA plans is greater than or equal to 75%.
Level of and change in physical activity levels | 12 weeks
  The mean number of Metabolic Equivalent Task (MET) hours per week that participants engaged in physical activity as well as the number of minutes per week that participants engaged in light, moderate, and vigorous intensity PA for each of the experimental and control groups will be calculated.
Level of adherence to physical activity intervention | 12 weeks
  The number of weeks that each participant missed receiving the intervention will be calculated. In addition, qualitative data will be collected to assess the pattern of missed weeks for each participant including the reasons that any weeks were missed.
Level of adherence to intervention delivery | 12 weeks
  An intervention fidelity audit will be conducted. The percentage of audited participants that engaged in each of the main components of intervention delivery (i.e pre-baseline home visit, baseline home visit, and weekly telephone calls) will be calculated. In addition, the percentage of individual intervention delivery criteria items that were met in each component will be calculated for each audited participant.

SECONDARY OUTCOMES:
Caregivers' perception of the acceptability of the intervention | 12 weeks
  Qualitative data will be collected during the weekly telephone calls and follow-up interviews to evaluate the acceptability of the structure, content, and process of the physical activity intervention.
  This criterion for advancing to a full RCT will be met if <10% of participants report major complaints about the intervention.
Caregivers' perception of benefits and/or risks of intervention | 12 weeks
  Qualitative data will be collected at the follow-up interviews to determine caregivers' overall perception of whether or not and in what ways the physical activity intervention impacted them.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Penner, RN, PhD(c), Principal Investigator — McGill University; Jewish General Hospital; S Robin Cohen, PhD, Principal Investigator — McGill University; Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada